CLINICAL TRIAL: NCT07209566
Title: The Effect of Vaginal Somatovisceral Pain on Hip Extension Mobility and Strength in Women at Mid-cycle With Dysmenorrhea vs. Controls: A Case-control Study
Brief Title: A Research Study Exploring How Musculoskeletal Function and the Autonomic Nervous System Relate to Visceral Pain in Women With and Without Dysmenorrhea (Painful Periods).
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azusa Pacific University (Other)
Responsible Party: Principal Investigator, Megan Steele, PhD candidate, Azusa Pacific University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-116
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Dysmenorrhea; Dysmenorrhea Primary; Visceral Pain; Menstrual Pain
Keywords: Effect of visceral organ pain on musculoskeletal and autonomic nervous system
MeSH Terms: conditions — Dysmenorrhea; Visceral Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visceral Pain Stimulus (Experimental): All participants will receive a visceral pain stimulus and have their hip range of motion and strength tested before and after the stimulus. Their heart rate variability will be measured throughout.
  Interventions: Diagnostic Test: Visceral Pain Stimulus

INTERVENTIONS:
Diagnostic Test: Visceral Pain Stimulus — Participants will receive a visceral pain stimulus while being monitored for heart rate variability (HRV), and will have hip mobility and dorsiflexor strength assessed before and after.

SUMMARY:
The purpose of this clinical trial is to determine if women with dysmenorrhea demonstrate an increased musculoskeletal and autonomic nervous system response to a painful visceral stimulus compared to controls. A secondary aim is to determine if interoceptive awareness moderates this relationship. The designed methodology aims to elucidate the intricate connections between the interoceptive and musculoskeletal systems in pain perception among female participants, providing valuable insights into the underlying mechanisms of interoceptive pain and functional musculoskeletal changes.

DETAILED DESCRIPTION:
A case-control trial will be conducted. The experimental group will consist of at least 30 subjects with a pain rating during menstruation greater than or equal to 4. The control group will be age-matched participants with pain rating less than or equal to 3 during menstruation. The study will consist of one information and instrumentation session followed by one lab session. During the initial session, participants will fill out demographic information and the VAS to allow for stratification into experimental or control groups. They will be given an LH test kit and educated on how to perform LH tests. They will be asked to track their menstrual cycle on an app or online journal that can be shared with investigators. They will be asked to download an HRV app and be taught how to measure their HRV using their phone's camera. They will be instructed to take a one-minute measure of HRV once daily for 30 days beginning on the first day of their period.

On lab day, participants will be asked to remove clothing and put on a gown, booties, and disposable underwear to wear during testing. They will be led into a temperature-controlled environment where they will complete the testing. Testing includes HRV baseline measurement for 5 minutes, heartbeat counting for 3 short sessions (25, 35, and 45 seconds), and confidence about scoring. Next, an investigator with a certification to complete internal pelvic exams will ask the participant to lie on the table, and a student investigator will take the baseline measurement of their hip extension. The side being measured will be randomized, and only one side will be tested on each participant.

Next, the barostat probe will be inserted into the vaginal canal. The barostat will be inflated once to allow the participant to experience the sensation of the balloon. The probe will then be inflated until the participant reports the sensation of pain. The amount of distension in the balloon will be recorded, and hip mobility will again be measured. The purpose of this clinical trial is to determine if women with dysmenorrhea demonstrate an increased musculoskeletal and autonomic nervous system response to a painful visceral stimulus compared to controls.

ELIGIBILITY:
Inclusion Criteria: Non-pregnant women, not taking hormonal birth control, between the ages of 18 and 36 who report regular menstrual cycles are eligible for the study Exclusion Criteria: Participants will be excluded if they are currently pregnant or, have given birth within the preceding six months, are breastfeeding, or are undergoing in-vitro fertilization treatments. Exclusions also include those who have had abdominal, lumbar, or pelvic surgery within the preceding 12 months, suffer from a chronic pain condition, have an active genitourinary infection, are incontinent of bowel or bladder, or have been diagnosed with prolapse of a pelvic organ, severe labral pathology, femoral acetabular impingement (FAI), interstitial cystitis, endometriosis, pelvic inflammatory disease, irritable bowel syndrome, or other pelvic pathology. Participants reporting a cycle length of less than 28 days or longer than 35 days, those with a history of sexual assault, and those who are anovulatory without hormonal BC or amenorrheic will also be excluded.

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women are eligible for this study because it requires a vaginal canal and a uterus.
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in hip range of motion | Change from baseline to immediately after the pain stimulus is given.
  The change in hip range of motion from baseline to after a visceral pain stimulus is a primary outcome measure of this study. This measurement will be compared between groups to determine if those with dysmenorrhea react to a painful stimulus differently compared to those without dysmenorrhea.
Change in dorsiflexor strength | From baseline to immediately after the pain stimulus.
  The change in strength of ankle dorsiflexors on the contralateral side of the hip being measured will also be assessed. This will be measured before and after the visceral pain stimulus to determine if there is a change. This measurement will be compared between groups to determine if those with dysmenorrhea react to a painful stimulus differently compared to those without dysmenorrhea.
Heart Rate Variability | From baseline to the end of the lab testing session, approximately 60 minutes.
  Heart rate variability will be measured throughout, and several time frames will be marked, including a 5-minute baseline within a 15-minute session, at the time of insertion of the probe, and at the pain stimulus, to determine if those with dysmenorrhea react to a painful stimulus differently compared to those without dysmenorrhea.

SECONDARY OUTCOMES:
Interoceptive awareness | During the testing day, following physical pain stimulus.
  Participants will also be given the multidimensional analysis of interoceptive awareness, 2nd edition (MAIA-2), to assess their interoceptive awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Derrick Sueki, PT, PhD, DPT, Study Chair — Azusa Pacific University
Locations (1):
- Azusa Pacific University, Azusa, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared to protect confidentiality.

REFERENCES:
- [Background] Pacheco-Carroza EA. Visceral pain, mechanisms, and implications in musculoskeletal clinical practice. Med Hypotheses. 2021 Aug;153:110624. doi: 10.1016/j.mehy.2021.110624. Epub 2021 Jun 6. PMID 34126503
- [Background] Serrano-Imedio A, Calvo-Lobo C, Casanas-Martin C, Garrido-Marin A, Pecos-Martin D. Myofascial Pain Syndrome in Women with Primary Dysmenorrhea: A Case-Control Study. Diagnostics (Basel). 2022 Nov 7;12(11):2723. doi: 10.3390/diagnostics12112723. PMID 36359567
- [Background] Tu FF, Epstein AE, Pozolo KE, Sexton DL, Melnyk AI, Hellman KM. A noninvasive bladder sensory test supports a role for dysmenorrhea increasing bladder noxious mechanosensitivity. Clin J Pain. 2013 Oct;29(10):883-90. doi: 10.1097/AJP.0b013e31827a71a3. PMID 23370073
- [Background] Tucker K, Larsson AK, Oknelid S, Hodges P. Similar alteration of motor unit recruitment strategies during the anticipation and experience of pain. Pain. 2012 Mar;153(3):636-643. doi: 10.1016/j.pain.2011.11.024. Epub 2011 Dec 29. PMID 22209423
- [Background] Van Oudenhove L, Kragel PA, Dupont P, Ly HG, Pazmany E, Enzlin P, Rubio A, Delon-Martin C, Bonaz B, Aziz Q, Tack J, Fukudo S, Kano M, Wager TD. Common and distinct neural representations of aversive somatic and visceral stimulation in healthy individuals. Nat Commun. 2020 Nov 23;11(1):5939. doi: 10.1038/s41467-020-19688-8. PMID 33230131
- [Background] Yacubovich Y, Cohen N, Tene L, Kalichman L. The prevalence of primary dysmenorrhea among students and its association with musculoskeletal and myofascial pain. J Bodyw Mov Ther. 2019 Oct;23(4):785-791. doi: 10.1016/j.jbmt.2019.05.006. Epub 2019 May 14. PMID 31733762
- [Background] Wakefield CB, Halls A, Difilippo N, Cottrell GT. Reliability of goniometric and trigonometric techniques for measuring hip-extension range of motion using the modified Thomas test. J Athl Train. 2015 May;50(5):460-6. doi: 10.4085/1062-6050-50.2.05. Epub 2015 Jan 6. PMID 25562458

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT07209566/Prot_SAP_000.pdf